CLINICAL TRIAL: NCT06943040
Title: Validity and Reliability of 6-minute Pegboard and Ring Test in Individuals With Spinal Cord Injury
Brief Title: Validity and Reliability of 6-minute Pegboard and Ring Test
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, PhD, Istinye University
Other Study IDs: 1111
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; 6PBRT; Validity; Reliability
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Other: There will be no intervention on the participants within the scope of this study.

INTERVENTIONS:
Other: There will be no intervention on the participants within the scope of this study. — There will be no intervention on the participants within the scope of this study.

SUMMARY:
Spinal Cord Injury (SCI) is a severe neurological condition that occurs as a result of traumatic or non-traumatic causes and results in motor, sensory, and/or autonomic dysfunction. The daily life of individuals with SCI often consists of low activity levels, which can cause loss of physical condition. Therefore, the participation of individuals with SCI in exercise is necessary to improve cardiovascular health and function, as well as to increase life expectancy and quality. Determining the strength, endurance, and exercise capacity of the upper extremities in individuals with SCI is an important issue in the management of SCI. One of the tests that serves this purpose is the six-minute pegboard and ring test (6PBRT). Since 6PBRT is used in clinical and research applications in individuals with SCI, it is important to know its validity and reliability. This study aims to investigate the validity and reliability of 6PBRT in individuals with SCI.

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) is a severe neurological condition that occurs as a result of traumatic or non-traumatic causes and results in motor, sensory, and/or autonomic dysfunction. Serious and long-term social, physical, and psychological problems that occur following the injury, a rapid decrease in the quality of life of patients, and economic problems such as loss of employment make SCI an important problem with both individual and societal dimensions. The annual SCI incidence is 12.7/million in our country, and the average age of injury is 35.5.

Secondary complications that occur in the short and long term following SCI play an important role in the continuity of care of individuals with SCI. According to the data of the National SCI Statistics Center (NSCISC), complications such as pneumonia, atelectasis, deep vein thrombosis, pulmonary embolism, pressure ulcers, autonomic dysreflexia, renal problems, and fractures are very common after SCI. It is thought that these complications resulting from SCI are a direct result of immobility. In addition, physical inactivity causes loss of functional independence, decreases quality of life, and significantly affects social participation. The daily life of individuals with SCI often consists of low activity levels and leads loss of physical condition. Therefore, the participation of individuals with SCI in exercise and improvement of cardiovascular health and function is necessary to increase life expectancy and quality. Various upper extremity exercises have been shown to improve the general condition of individuals with SCI. Determination of upper extremity strength, endurance, and exercise capacity in individuals with SCI is an important issue in the management of SCI. One of the tests that serves this purpose is the six-minute pegboard and ring test (6PBRT), which is valid and reliable in individuals with chronic obstructive pulmonary disease. Since 6PBRT is used in clinical and research applications in individuals with SCI, it is important to know its validity and reliability. This study aims to investigate the validity and reliability of 6PBRT in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* At least one year since the spinal cord injury
* Being an adult (≥18 years old)
* Injury level between T1 and L5
* Being a full-time wheelchair (WD) user for mobility

Exclusion Criteria:

- Have additional medical conditions (upper extremity and shoulder injuries, etc.) that may affect their ability to perform the tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals With Spinal Cord Injury
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
6-minute pegboard and ring test | 1 week
  The 6PBRT is an upper extremity exercise test that evaluates upper extremity functional capacity through unsupported arm activities. The 6PBRT apparatus consists of four bars placed horizontally on the wall, two at shoulder height and the other two 20 centimeters (cm) above shoulder height. Initially, 10 rings are placed on the lower two bars. Participants sit in a chair in front of the apparatus with back support and feet in full contact with the floor. Participants are instructed to move two rings at a time from the lower bar to the upper bar with both hands (one on each side). When 20 rings are placed from the lower bars to the upper levels, participants are asked to return the rings to the lower level. This sequence of movements is repeated for six minutes. The number of rings moved during the test is used as the final score representing performance. Participants are verbally encouraged every minute during the test, and the verbal command is standardized.
Shoulder flexor muscle strength | 1 week
  Muscle strength will be measured using a digital dynamometer with the patient in a sitting position. Muscle tests will be repeated three times for each side, and the highest value will be recorded in kg.
Shoulder abductor muscle strength | 1 week
  Muscle strength will be measured using a digital dynamometer with the patient in a sitting position. Muscle tests will be repeated three times for each side, and the highest value will be recorded in kg.
Elbow extensor muscle strength | 1 week
  Muscle strength will be measured using a digital dynamometer with the patient in a sitting position. Muscle tests will be repeated three times for each side, and the highest value will be recorded in kg.
Elbow flexor muscle strength | 1 week
  Muscle strength will be measured using a digital dynamometer with the patient in a sitting position. Muscle tests will be repeated three times for each side, and the highest value will be recorded in kg.
Handgrip strength | 1 week
  The participant will be measured using a hand dynamometer in a sitting position. Muscle tests will be repeated three times for each side, and the highest value will be recorded in kg.
The 20-m propulsion test (MWPT 20m ) | 1 week
  It will be used to evaluate the participants' ability to use a manual wheelchair. A 20-meter track was set up by drawing a line at the beginning and end. Patients were asked to drive their wheelchairs as fast as they could on this 20-meter track. During this time, the evaluator determined how many seconds it took to complete the 20-meter track with a stopwatch, and the results were recorded in seconds.
Modified Functional Reach Test (mFUT) | 1 week
  This test is a quick and easy-to-use test that can be used to measure sitting balance in individuals with SCI. The test is performed while the patient is sitting in a wheelchair with their hips, knees, and ankles flexed at 90 degrees. Individuals place their upper extremities at 90 degrees of flexion in the starting position. After measuring with an inflexible tape measure in this position, patients extend as far as they can and measure again. The distance between them is measured and recorded in centimeters. Participants performed flexion and abduction extensions for the right and left upper extremities separately, and the results will be recorded in centimeters (cm).

SECONDARY OUTCOMES:
Barthel Index (BI) | 1 week
  BI is a scale that evaluates all steps of daily living activities. It is used to determine the level of independence of individuals in their activities. The scores of the Barthel index vary between 0-100, 0-20 points; completely dependent, 21-61 points; advanced dependent, 62-90 points; moderate dependent, 91-99 points; mild dependent, 100 points; independence.